CLINICAL TRIAL: NCT03420300
Title: Elbasvir/Grazoprevir for Treatment-naive and Treatment-experienced Patients With Hepatitis C Virus Genotype 1b Receiving Hemodialysis
Brief Title: EBR/GZR for HCV-1b Patients Receiving Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201709053MIPC
Record Dates: First submitted 2018-01-28; First posted 2018-02-05 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C virus; Hemodialysis; Direct acting antiviral agent
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBR/GZR (Experimental): Elbasvir/grazoprevir (EBR/GZR 50mg/100mg fixed dose combination [FDC]): 1 table per os per day for 12 weeks
  Interventions: Drug: EBR/GZR

INTERVENTIONS:
Drug: EBR/GZR — Elbasvir/grazoprevir (EBR/GZR 50mg/100mg fixed dose combination [FDC]): 1 table per os per day for 12 weeks
  Other Names: Zepatier

SUMMARY:
Hepatitis C virus (HCV) infection is common in patients receiving hemodialysis. The uptake of antiviral therapy for these patients is limited in the era of interferon (IFN) plus ribavirin (RBV), probably because the sustained virologic response (SVR) rates are low and the risk of treatment-related adverse events (AEs) are high. In the era of IFN-free direct acting antiviral agents (DAAs), several studies have indicated high rates of SVR and excellent safety profiles to treat patients with severe renal impairment. With regard to elbasvir/grazoprevir (EBR/GZR) treatment, a phase 3 study (C-SURFER) study has shown 99% of SVR in HCV-1 patients with chronic kidney disease (CKD) stage 4 or 5. Furthermore, most patients tolerated the treatment well. Although the data confirmed the excellent safety and efficacy in HCV-1 patients with severe renal impairment, data regarding the safety and efficacy for Asian HCV-1b patients receiving hemodialysis is lacking. Therefore, we aim to evaluated the safety and efficacy of EBR/GZR for 12 weeks in treatment-naive and treatment-experienced HCV-1b patients receiving hemodialysis.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection remains a major co-morbidity in hemodialysis patients. The incidence and prevalence rates of HCV infection in hemodialysis patients are much higher than those in the general population, and are attributed to high rates of nosocomial HCV transmission. With regard to HCV genotype distribution, HCV genotype 1 (GT-1) infection is the most prevalent type of infection worldwide and the genotype distribution in HCV-infected individuals receiving hemodialysis (HD) is similar to that observed in HCV-infected individuals with normal renal function. Compared to non-HCV infected hemodialysis patients, HCV-infected patients have increased risks of liver-related morbidity and mortality. Although HCV-infected hemodialysis patients who receive renal transplantation have survival advantages over those who remain on maintenance dialysis, these patients still have poor patient and graft survival, as well as have poor responses to interferon (IFN)-based therapy.In contrast, hemodialysis patients who eradicate HCV infection have improved biochemical, virologic and histologic responses, whether on maintenance dialysis or after renal transplantation.

Approximately one third of hemodialysis patients with chronic HCV infection achieve sustained virological response (SVR) by conventional IFN or peginterferon monotherapy.In addition 18-30% of patients receiving IFN-based monotherapy prematurely discontinued treatment due to adverse events (AEs). Although the addition of ribavirin to IFN further improves the SVR rate in HCV-infected patients with normal renal function, ribavirin has been considered contraindicated to treat HCV-infected hemodialysis patients because of concern for life-threatening hemolytic anemia. Recently, pilot studies have indicated the feasibility of adding low-dose ribavirin (200 mg three times per week to daily 400 mg, adjusted to achieve a target concentration of 10-15 μmol/L), to IFN for treatment of HCV-infected hemodialysis patients. Generally, the SVR rate and the premature discontinuation rate due to null-response, severe anemia, and/or heart failure for combination therapy are 56% and 22%, respectively. Based on these small-scale studies, low-dose ribavirin (daily 200 mg) was approved in August 2011 by the U.S. Food and Drug Administration to treat HCV-infected hemodialysis patients.30 Two recent well-conducted randomized control studies to compare the efficacy and safety of combination therapy with peginterferon alfa-2a (135 μg/week) plus low-dose ribavirin (RBV) (200 mg/day) or monotherapy with peginterferon (135 μg/week) for 48 and 24 weeks in treatment-naïve HCV GT-1 and GT-2 infected individuals receiving hemodialysis showed that the SVR rates of combination therapy groups were greater than those of monotherapy groups (64% versus 34%, p < 0.001 for HCV GT-1; 74% versus 44%, p < 0.001 for HCV GT-2), respectively. Although the SVR rate of combination therapy with peginterferon plus low-dose ribavirin is higher than that of peginterferon monotherapy. About 70-75% of these patients experienced clinically significant anemia which needed high dose of erythropoiesis stimulating agents (ESAs) to keep the hemoglobin level within the safety range. Although telaprevir (TVR)-based triple therapy has been used to treat 4 HCV-1 patients receiving hemodialysis who were not responsive to prior peginterferon plus RBV with good efficacy, the added on-treatment adverse events (AEs) and the pill burden precluded the widespread use of this agent.

The recent introduction of IFN-free direct acting antiviral agents (DAAs) has made a paradigm shift with regard to the medical treatment for HCV-infected individuals, based on the excellent efficacy and safety in ordinary patients. Among the various IFN-free DAA regimens, treatment with elbasvir/grazoprevir (EBR/GZR) has been approved in 2016 to treat patients with chronic HCV GT-1 and GT-4 infection. Treatment with EBR/GZR with/without weight-based ribavirin for 12-16 weeks achieved an SVR12 rate of 94-100% in treatment-naïve and PR or protease-inhibitor based treatment-experienced HCV GT-1a, GT-1b or GT-4 patients, respectively (C-EDGE TN, TE, SALVAGE). Furthermore, the SVR12 rates in HIV-coinfected patients with HCV GT-1a, GT-1b and GT-4 were 95.3% and 98.0% by using EBR/GZR for 12 weeks (C-EDGE Coinfection). In addition to high SVR rates by 12-16 weeks of EBR/GZR treatment, the overall safety profiles are excellent, with only 1% of the patients who discontinue treatment due to drug-related adverse event. With regard to constitutional symptoms, treatment with EBR/GZR had comparable rates to the placebo arms. With regard to laboratory abnormalities, about 1% and less than 1% of the treatment patients experience AST/ALT elevation and hyperbilirubinemia. Clinically significant anemia is more commonly encountered in patients receiving EBR/GZR with weight-based ribavirin. Taking together, treatment with EBR/GZR is efficacious and safe for HCV-infected subjects with HCV GT-1 or 4 infection. The post-hoc analyses for potential factors affecting the SVR rates showed that among GT-1a infected patients with baseline NS5A resistant associated variants (RAVs) at position of 28, 30, 31 and 93, the SVR rates will be compromised for those receiving 12 weeks of treatment or without adding RBV. In addition, treatment-experienced HCV GT-4 patients should also receive 16 weeks of EBR/GZR plus RBV to secure the SVR rates. In GT-1a or GT-1b patients who fail prior protease inhibitor-based triple therapy, 12 weeks of GZR/EBR plus RBV are recommended to secure the high SVR rates. For GT-1a treatment-naïve or PR-experienced patients without the presence of baseline NS5A RAVs, GT-1b treatment-naïve or PR-experienced patients or GT-4 treatment-naïve patients, EBR/GZR for 12 weeks offer satisfactory safety and efficacy profiles. Gender, ethnicity, age, interleukin-28B (IL28B) genotype, cirrhosis status and baseline HCV RNA levels do not affect the overall SVR rates in EBR/GZR treatment patients.

The pharmacokinetic (PK) study of elbasvir and grazoprevir was evaluated 16 subjects with severe renal impairment and end-stage renal disease (ESRD) on maintenance hemodialysis and matched healthy controls. Compared to subjects with matched healthy controls, the area under the curves (AUCs) of elbasvir in subjects with severe renal impairment and ESRD were 99% and 86%; the AUCs of grazoprevir in subjects with severe renal impairment and ESRD were 85% and 83%, respectively. The pharmacokinetic study indicated that dose dosage adjustments of EBR/GZR are not needed for patients with severe renal impairment or those who are on maintenance hemodialysis.

The phase 3 C-SUFER study evaluated the safety and efficacy of EBR/GZR BV for 12 weeks in a total of 235 treatment-naïve and treatment-experienced HCV GT-1 patients with severe renal impairment or ESRD.42 About 82% of the patients had chronic kidney disease (CKD) stage 5, and the remaining 18% of the patients had CKD stage 4. The full set and the modified full set analyses for SVR12 in patients receiving 12 weeks of treatment were 94% and 99% respectively. On-treatment undetectable HCV RNA levels at weeks 4 and 12 were 90% and 100%, respectively. In patients with ESRD, the overall SVR12 was 98.9%. No patients discontinued the study drugs due to adverse events. Furthermore, the constitutional and the laboratory abnormalities were mild in grades and were lower in frequency, compared to the control arm. This large-scale study shows that treatment with EBR/GZR is efficacious and safe for HCV-1 patients with severe renal impairment and those with end-stage renal disease.

Although peginterferon monotherapy and combination therapy with peginterferon plus low-dose RBV for 24-48 weeks have been evaluated in many studies, the efficacy for the treatment regimens were only modest (SVR rate about 60%). In addition, the on-treatment AEs and SAEs by IFN-based therapies were frequently encountered in HCV-infected patients receiving hemodialysis. Of note was the pronounced on-treatment hemoglobin level decrease in patients receiving combination therapy by peginterferon plus low-dose RBV, necessitating significant RBV dose reduction and high-dose erythrocyte stimulating agent (ESA) support.

By receiving IFN-free DAA therapies, HCV-infected patients have excellent SVR rates, low on-treatment SAE and AE rates, shorter treatment duration, and low pill burdens. The PK study of EBR/GZR proves the excellent safety profiles and dose adjustment are not needed for EBR/GZR regimen in subjects with various degrees of renal impairment. The C-SURFER study showed the excellent on-treatment and off-therapy antiviral effects in HCV GT-1a and GT-1b infected patients receiving EBR/GZR, respectively. However, the C-SURFER study enrolled only limited patients of Asian ancestry, making the safety and efficacy in this group of patients still to be confirmed. Based on the excellent safety and efficacy profiles of EBR/GZR treatment for HCV GT-1b infected patients with normal renal function, we aim to evaluate the safety and efficacy of EBR/GZR for 12 weeks in treatment-naïve and treatment-experienced HCV GT-1b patients receiving hemodialysis in Asian population, taking HCV GT-1b patients treated by peginterferon plus ribavirin for 48 weeks as the historical control.

ELIGIBILITY:
Inclusion Criteria:

* 20 yeas or more
* Male or female
* Body mass index (BMI) 18.5-35.0 kg/m2
* Chronic HCV infection, defined as patients who meet as least one of the two following criteria:

  1. Anti-HCV antibody (Abbott HCV EIA 2.0, Abbott Laboratories, Abbott Park, Illinois, USA) or HCV RNA > 1,000 IU/mL for at least 6 months before screening
  2. Positive HCV RNA > 1,0000 IU/mL (Cobas TaqMan HCV Test v2.0, Roche Diagnostics GmbH, Mannheim, Germany, low limit of quantification (LLOQ): 25 IU/mL) at the time of screening with a liver biopsy consistent with chronic HCV infection
* HCV genotype 1 (HCV GT-1b) infection (Abbott RealTime HCV genotype II, Abbott Molecular Inc. Illinois, USA)
* Treatment-naïve or treatment-experienced (including patients who relapsed, who had virological breakthrough, or who were null-responsive to IFN-based therapies)
* HCV RNA > 10,000 IU/mL at screening
* Estimated glomerular filtration (eGFR) rate < 15 mL/min/1.73m2 as assessed by modified of diet in renal disease (MDRD) equation, and receiving regular hemodialysis

Exclusion Criteria:

* HCV infection other than HCV GT-1b
* HBV or HIV coinfection
* Presence of decompensated cirrhosis (Child-Pugh class B or C)
* Any primary cause of liver disease other than chronic HCV infection, including but not limited to the following

  1. Hemochromatosis
  2. Alfa-1 antitrypsin deficiency
  3. Wilson's disease
  4. Autoimmune hepatitis
  5. Alcoholic liver disease
  6. Drug-induced hepatitis
  7. Screening laboratory analyses showing any of the following results

     * Hemoglobin (Hb) level < 10 g/dL
     * Absolute neutrophil count (ANC) < 1,500 cells/μL
     * Platelet count < 70,000 cells/mm3
     * International normalized ratio (INR) > 2.0
     * Albumin (Alb)< 3.0 g/dL
     * Bilirubin (Bil) > 2.0 mg/dL
     * Alanine aminotransferase (ALT) > 10X upper limit of normal (ULN)
     * Aspartate aminotransferase (AST) > 10X upper limit of normal (ULN)
     * Serum alfa-fetoprotein (AFP) > 100 ng/mL
* Presence of hepatocellular carcinoma (HCC) on imaging studies such as computed tomography (CT) scan or magnetic resonance imaging (MRI)
* History of malignancy (except cutaneous melanoma) within 5 years at the screening
* Organ transplantation other than cornea and hair (prior renal transplantation with graft failure not included)
* Prior exposure to investigational agents for HCV (direct acting antiviral agents, host-targeting agents, or therapeutic vaccines)
* Pregnancy
* Unwilling to have contraception during the study period
* Unwilling to provide informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2020-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, PhD, Study Director — National Taiwan University Hospital
Locations (6):
- Taiwan (6):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University, Taipei
  - Far Eastern Memorial Hospital, Taipei County

IPD SHARING:
Plan to Share IPD: No
Confidential of the individual participant data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 medical center in Taiwan to evaluate the tolerability and efficacy of elbasvir/grazoprevir (EBR/GZR) for patients with hepatitis C virus genotype 1 infection and receiving hemodialysis. The recruitment period was from 05 June, 2018 to 30 April, 2019
Pre-assignment Details: The study was an one-arm, open label, multi-center study. Patients were checked for inclusion and exclusion criteria to assess the eligibility. There was no pre-assignment criteria in the study.
Period: Overall Study
Arm/Group | EBR/GZR
Started | 40
Completed | 38
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | EBR/GZR
Number analyzed (Participants) | 40
Age, Customized [Median (Full Range); unit: years] | 64 [32 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 40
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 40
Treatment-naive [Count of Participants; unit: Participants] | 35
History of renal transplantation [Count of Participants; unit: Participants] | 5
Diabetes mellitus [Count of Participants; unit: Participants] | 13
Hypertension [Count of Participants; unit: Participants] | 23
Dyslipidemia [Count of Participants; unit: Participants] | 8
Hemoglobin [Median (Full Range); unit: g/dL] | 11.8 [10.1 to 14.8]
Absolute neutrophil count [Median (Full Range); unit: 10^9 cells/L] | 3.7 [2.0 to 7.1]
Platelet count [Median (Full Range); unit: 10^9 cells/L] | 196 [100 to 345]
International normalized ratio (INR) [Median (Full Range); unit: ratio] | 1.01 [0.89 to 1.26]
Albumin [Median (Full Range); unit: g/dL] | 4.3 [3.5 to 5.1]
Total bilirubin [Median (Full Range); unit: mg/dL] | 0.5 [0.1 to 1.0]
Alanine aminotransferase [Median (Full Range); unit: IU/L] | 28 [8 to 156]
Creatinine [Median (Full Range); unit: mg/dL] | 7.3 [4.2 to 15.4]
eGFR [Median (Full Range); unit: mL/min/1.73m^2] | 7 [3 to 10]
IL28B rs2979860 non-CC genotype [Count of Participants; unit: Participants] | 6
HCV RNA [Median (Full Range); unit: Log10 IU/mL] | 5.60 [4.18 to 7.28]
HCV RNA > 800,000 IU/mL [Count of Participants; unit: Participants] | 11
Liver stiffness measurement (LSM) [Median (Full Range); unit: kPa] | 7.1 [3.3 to 57.9]
Fibrosis stage [Count of Participants; unit: Participants] — Liver stiffness measurement (LSM, Fibroscan) for fibrosis staging
  1. F0-1 (minimal or no fibrosis): < 7.0 kPa (kiloPascal)
  2. F2 (significant fibrosis): 7.1-9.4 kPa (kiloPascal)
  3. F3 (advanced fibrosis): 9.5-12.3 kPa (kiloPascal)
  4. F4 (cirrhosis): > or = 12.4 kPa (kiloPascal)
  Participants
    F0-1 | 20
    F2 | 14
    F3 | 2
    F4 | 4
Resistance associate substitution (RAS) [Count of Participants; unit: Participants]
  NS3 | 33
  NS5A | 7

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR12) Rate
Description: Proportion of patients who had undetectable serum HCV RNA 12 weeks after the completion of elbasvir/grazoprevir (EBR/GZR)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | EBR/GZR
Number analyzed (Participants) | 40
Participants | 38

2. Secondary Outcome: Treatment-emergent Adverse Event (AE)-Related Withdrawal Rate
Description: Proportion of participants who withdrew from the study due to any adverse events (AEs) which were judged related to elbasvir/grazoprevir (EBR/GZR)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | EBR/GZR
Number analyzed (Participants) | 40
Participants | 0

3. Secondary Outcome: Sustained Virologic Response (SVR24) Rate
Description: Proportion of patients who had undetectable serum HCV RNA 24 weeks after the completion of elbasvir/grazoprevir (EBR/GZR)
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | EBR/GZR
Number analyzed (Participants) | 40
Participants | 38

4. Secondary Outcome: Rapid Virologic Response (RVR) Rate
Description: Proportion of patients who had undetectable serum HCV RNA at week 4 of elbasvir/grazoprevir (EBR/GZR) treatment
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | EBR/GZR
Number analyzed (Participants) | 40
Participants | 39

5. Secondary Outcome: End-of-treatment Virological Response (EOTVR) Rate
Description: Proportion of patients who had undetectable serum HCV RNA at the time point of treatment completion for elbasvir/grazoprevir (EBR/GZR)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | EBR/GZR
Number analyzed (Participants) | 40
Participants | 40

6. Secondary Outcome: Week 12 Virologic Response (W12VR)
Description: Proportion of patients who completed 12 weeks of elbasvir/grazoprevir (EBR/GZR) treatment and who had undetectable serum HCV RNA at week 12 of treatment
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | EBR/GZR
Number analyzed (Participants) | 40
Participants | 39

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | EBR/GZR
All-Cause Mortality (participants affected / at risk) | 2/40
Serious Adverse Events (participants affected / at risk) | 5/40
Other Adverse Events (participants affected / at risk) | 7/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBR/GZR (N=40)
Suicide (General disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac arrrythmia (Cardiac disorders) | 1 (1)
Non-variceal gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Hepatocellular carcinoma (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBR/GZR (N=40)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This study enrolled the tolerability and efficacy in East-Asian patients, where the results may not be generalized to other races.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03420300/Prot_SAP_000.pdf